CLINICAL TRIAL: NCT01542515
Title: Allograft Meniscal Arthroplasty for the Treatment of Basal Joint Arthritis of the Thumb
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Collaborators: LifeNet Health (Industry)
Responsible Party: Principal Investigator, Paul S. Shapiro, M.D., Paul S. Shapiro, M.D., Corewell Health East
Other Study IDs: 2008-298
Record Dates: First submitted 2012-02-24; First posted 2012-03-02 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Arthritis
Keywords: Allograft; Arthroplasty; Basal Joint; carpometacarpal joint; Thumb; meniscus; osteoarthritis; Patients with Stages I - III arthritis of the the thumb carpometacarpal joint
MeSH Terms: conditions — Arthritis; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Osteoarthritis of the carpometacarpal joint of the thumb: The group of patients enrolled in this study all have the diagnosis of carpometacarpal arthritis of the thumb. The patients did not respond favorably to non-operative management including oral anti-inflammatory medications, corticosteroid injections, and thumb splinting. Operative management was therefore recommended using the technique of meniscal allograft arthroplasty.
  Interventions: Procedure: Meniscal allograft arthroplasty of the carpometacarpal joint of the thumb

INTERVENTIONS:
Procedure: Meniscal allograft arthroplasty of the carpometacarpal joint of the thumb — The surgical procedure will involve the use of human meniscal allograft tissue that will be provided by industry. The meniscus will be contoured into a "T" shape. The T-shaped meniscus allograft is then inserted into the arthritic thumb CMC joint and secured with two suture anchors.

SUMMARY:
Hypothesis:

The use of knee meniscal allograft as a joint spacer and stabilizer is a viable option for the surgical treatment of basal joint arthritis of the thumb.

A variety of surgical procedures have been developed for the treatment of basal joint osteoarthritis of the thumb. Problems with persistent pain and poor function have been reported to some degree for each of these procedures. Using the concept of an implant acting as a spacer and stabilizer the investigators proposed and implemented a novel surgical technique using allograft knee meniscus as a biologic implant for the treatment of basal joint arthritis of the thumb.

DETAILED DESCRIPTION:
Hypothesis:

The use of knee meniscal allograft as a joint spacer and stabilizer is a viable option for the surgical treatment of basal joint arthritis of the thumb.

Introduction:

A variety of surgical procedures have been developed for the treatment of basal joint osteoarthritis of the thumb. Problems with persistent pain and poor function have been reported to some degree for each of these procedures. Promising results were originally reported (2004) for the Artelon carpometacarpal (CMC) implant (Small Bone Innovations, Morrisville, PA) procedure which utilized the concept of a spacer and stabilizer of the CMC joint . Recent studies however, have demonstrated problems due to a foreign body reaction with the Artelon implant requiring revision surgery. Using the concept of an implant acting as a spacer and stabilizer we proposed and implemented the use of allograft knee meniscus as a biologic implant in the treatment of basal joint arthritis of the thumb

Methods:

A prospective study was performed on four thumbs using an allograft knee meniscus transplanted into the thumb CMC joint using the surgical technique described for that of the Artelon implant (Small Bone Innovations, Morrisville, PA). Data collected included: pain level, grip strength, tip, key and pinch strength, carpometacarpal, metacarpophalangeal, interphalangeal, and oppositional range of motion, as well as Disabilities of the Arm, Shoulder, and Hand (DASH) scores. Interval radiographic analysis is to be performed. Endpoints for data collection will be at three months, six months, one, two, three, four, and five years follow up.

ELIGIBILITY:
Inclusion Criteria:

* Stage I - III osteoarthritis / traumatic arthritis of the thumb.

Exclusion Criteria:

* Exclusion criteria were diabetes mellitus, kidney insufficiency, OA in the STT joint, or malignancy within the past 10 years.

Ages: 25 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women of all ages having the diagnosis of osteoarthritis of the thumb.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2009-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) Score | 5 years
  The DASH Outcome Measure is a 30-item, self-report questionnaire designed to measure physical function and symptoms in people with any of several musculoskeletal disorders of the upper limb. The tool gives clinicians and researchers the advantage of having a single, reliable instrument that can be used to assess any or all joints in the upper extremity.

CONTACTS AND LOCATIONS:
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

REFERENCES:
- [Background] Nilsson A, Liljensten E, Bergstrom C, Sollerman C. Results from a degradable TMC joint Spacer (Artelon) compared with tendon arthroplasty. J Hand Surg Am. 2005 Mar;30(2):380-9. doi: 10.1016/j.jhsa.2004.12.001. PMID 15781363
- [Background] Hommen JP, Applegate GR, Del Pizzo W. Meniscus allograft transplantation: ten-year results of cryopreserved allografts. Arthroscopy. 2007 Apr;23(4):388-93. doi: 10.1016/j.arthro.2006.11.032. PMID 17418331